CLINICAL TRIAL: NCT01166594
Title: Use of Bevacizumab in Trabeculectomy Surgery. A Prospective, 2 Centre, Randomized, Controlled Trial
Brief Title: Use of Bevacizumab in Trabeculectomy Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Glaucoma Research Society of Canada (Other)
Responsible Party: Principal Investigator, Dr. Catherine Birt, MD, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 136783
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma; Optic Neuropathy; Fibrosis
Keywords: Glaucoma; Elevated Intraocular Pressure (IOP); Optic Neuropathy; Bleb Failure; Avastin (Bevacizumab)
MeSH Terms: conditions — Glaucoma; Optic Nerve Diseases; Fibrosis; Ocular Hypertension | interventions — Bevacizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab (Experimental): Tested Drug
  Interventions: Drug: Bevacizumab
- Control (Placebo Comparator): Control - BSS
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Bevacizumab — Intrableb injection
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Control — intrableb BSS injection
  Other Names: Saline
  Arms: Control

SUMMARY:
When a patient with glaucoma who has a pressure that is too high and causing damage to their vision, despite receiving the maximum amount of medication that can be tolerated, the decision is made to have glaucoma surgery. Trabeculectomy is the most common form of glaucoma surgery used to treat open angle glaucoma. During trabeculectomy, an opening is created in the eye and partially covered with a flap of tissue. This new opening allows fluid to drain out of the eye bypassing the clogged drainage channels that are malfunctioning in patients with glaucoma. Studies have found that trabeculectomy significantly reduces vision loss and lowers eye pressure.

However, many people need another trabeculectomy or other glaucoma surgery because the surgery may fail either early or much later because the body closes the drain created by the surgeon. The surgery is also less likely to work in patients with darker pigmentation, children who have congenital glaucoma, people with difficult to control glaucoma with new blood vessels growing on the iris, diabetes or persons with prior eye surgery. As a result, the investigators need to find ways to improve the longterm survival of trabeculectomy surgery in all patients.

DETAILED DESCRIPTION:
The usual treatment is to not have an injection of Bevacizumab on the third through fifth day after trabeculectomy surgery. Topical anaesthetic drops to numb the eye will be given, prior to being given the tested medicine. Once the eye has been anaesthetized, the medication will be injected into the potential space created during the glaucoma surgery, also called a bleb, using a standard small syringe. The patient will receive an injection of either 1.25mg (0.05ml) of Bevacizumab or Balanced Salt Solution (BSS) into the trabeculectomy bleb that had been created in the surgery. Participants will be randomly (by chance) placed in one of the 2 study groups. There will be a 50% chance of being placed in either group. There will be 60 people who will participate in this study at 2 centres throughout the Toronto region. The length of this study for participants is 12 months, and the entire study is expected to take about 18 months to complete.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Patients with glaucoma that is inadequately controlled on maximal tolerated medical therapy and scheduled for trabeculectomy surgery (with/without combined cataract extraction)
* Decision makers fluent in English
* Decision makers able to understand and read consent form

Exclusion Criteria:

* Patients with active intraocular inflammation/uveitis or neovascular glaucoma
* History of previous trabeculectomy surgery or prior retinal detachment with scleral buckle placement in the surgical eye
* Aphakia in surgical eye
* Pregnant and nursing women
* Unable to fulfill inclusion criteria
* Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Birt, MD, FRCSC, Principal Investigator — Sunnybrook Hospital
Locations (1):
- Sunnybrook Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Tested Drug
  Bevacizumab: Intrableb injection - 30 patients
- Control: Control - BSS
  Control: intrableb BSS injection - 29 patients
Period: Overall Study
Arm/Group | Bevacizumab | Control
Started | 30 | 29
Completed | 23 | 24
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Control | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.8) | 61.3 (10.4) | 62.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 9 | 13 | 22
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Intraocular pressure comparison between the two groups at one year following surgery. A window of ±14 days was allowed for the one-year visit
Time Frame: One year
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bevacizumab | Control
Number analyzed (Participants) | 23 | 24
mm Hg | 13.9 (4.5) | 13.2 (5.1)
Statistical Analysis 1: Comparison: Bevacizumab vs Control; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Improved Bleb Appearance
Description: Improved bleb appearance was formally graded according to the Indiana bleb-grading scheme at each visit.
  The scheme has 4 sections: height of the bleb (H) with a range of H0 (flat bleb) to H4 (high bleb), horizontal extent of the bleb with a range of E0 (less than 1 clock hour) to E3 (more than 4 clock hours), vascularity of the bleb with a range of V0 (avascular) to V4 (extensive vascularity), and siedel test ranging from S0 (no leak) to S2 (streaming leak within 5 seconds).
  Each section was individually scored. Ophthalmic photographs of the surgical site were taken with patient consent. The photographs only included a small portion of the eye and the patient cannot be identified by them.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Control
Number analyzed (Participants) | 23 | 24
Participants | 14 | 12

3. Secondary Outcome: The Number of Participants Who Received 5-Fluorouracil (5-FU) Injections
Description: The number of participants who needed 5-FU injections during the first post-operative year for additional would modulation will be compared between the two groups.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Control
Number analyzed (Participants) | 23 | 24
Participants | 13 | 7

ADVERSE EVENTS:
Arm/Group | Bevacizumab | Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 14/23 | 11/24
Other Adverse Events (participants affected / at risk) | 6/23 | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=23) | Control (N=24)
Bleb leak (Eye disorders) | 8 (8) | 7 (7)
Hypotony (Eye disorders) | 14 (14) | 11 (11)
Choroidal Detachment (Eye disorders) | 6 (6) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=23) | Control (N=24)
Other (Eye disorders) | 6 | 7 — Other Adverse events included suprachoroidal hemorrhage, corneal abrasion, hyphema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No